CLINICAL TRIAL: NCT01738958
Title: Effect of Lozenges Containing Probiotic Lactobacilli on Enamel Demineralization Assed by QLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Mette Kirstine Keller, Assistant Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-4-2012-096
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Caries Dentalis
Keywords: Probiotic bacteria; Caries dentalis; QLF

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Probiotic lactobacilli (Active Comparator): L. reuteri, two times a day for 6 weeks
  Interventions: Biological: L. retueri
- Placebo (Placebo Comparator): Placebo tablets, two times a day for 6 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: L. retueri — two tablets a day for 6 weeks
  Arms: Probiotic lactobacilli
Biological: Placebo
  Arms: Placebo

SUMMARY:
Clinical trials in children and adults have suggested that daily consumption of probiotic lactic acid bacteria can reduce caries risk and caries development in primary teeth in preschool and stop root caries in the elderly. However, it is not known whether probiotic bacteria can affect the increased porosity in young permanent teeth in children and adolescents with many cavities.

It can be difficult to measure the increased porosity of the enamel by tooth decay, but this can be done using quantitative laser fluorescence (QLF). The method is based on visible light with a wavelength of 370 nm, addressing enamel. This produces an image consisting of red and green color tones and the dominant color of the enamel is green. Increased porosity of the enamel, resulting in a reduction of the auto-fluorescence and the loss (or gain) of the mineral can be quantified by means of a corresponding software.

The purpose of this study is to investigate the effect of a daily supplement of probiotic lactic acid bacteria on the loss of mineral in enamel assessed with QLF. The null hypothesis is that the mineral content will not differ from baseline in either the test group or the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* two sites with white spot lesions in anterior teeth

Exclusion Criteria:

* antibiotic treatment within 2 months

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in enamel porosity | Baseine and 12 weeks
  Change in enamel porosity assed by QLF

CONTACTS AND LOCATIONS:
Locations (1):
- Ishøj kommunale tandpleje, Ishøj, Denmark